CLINICAL TRIAL: NCT02013882
Title: 1-1-12 Wash-in for Desflurane Low Flow Anesthesia
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Other Study IDs: HE561247
Record Dates: First submitted 2013-12-05; First posted 2013-12-17 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Anesthesia
Keywords: low flow anesthesia; wash-in; desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1-1-12 wash-in: wash-in using O2:N2O 1:1 L/min with desflurane 12%
  Interventions: Procedure: 1-1-12 wash-in

INTERVENTIONS:
Procedure: 1-1-12 wash-in — wash-in phase during start of low flow anesthesia

SUMMARY:
We propose a new wash-in technique for desflurane low flow anesthesia with fresh gas flow of O2:N2O 1:1 L/min with desfluraene 12%.

The objective of this study is to identify time to achieve alveolar concentration of desflurane at1, 2, 3, 4, 5 and 6%.

DETAILED DESCRIPTION:
The benefits of low flow anesthesia are economic, less pollution, more heat and humidity preservation but it requires appropriate wash-in phase. The current wash-in protocols are complicated and time consuming. We propose a new 1-1-12 desflurane wash-in protocol which is more simple and predictable.

The objective of this study is to identify time to achieve alveolar concentration of desflurane at 1, 2, 3, 4, 5 and 6% with 1-1-12 wash-in protocol.

All patients will receive iv propofol 2 mg/kg as induction agent and succinyl choline 1.5 mg/kg for intubation. Then the ventilation will be controlled to achieve end-tidal CO2 30-35 mmHg with O2:N2O 1:1 L/min with desflurane 12%. Time to achieve alveolar concentration of desflurane at 1, 2, 3, 4, 5 and 6% will be recorded and analyzed. After that, the concentration of desflurane and anesthetic technique will be adjusted to requirement of anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II
* age 18-64 years

Exclusion Criteria:

* BMI > 35
* contraindicated for N2O
* with pulmonary or cardiac disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients undergoing general anesthesia with endotracheal intubation and controlled ventilation
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time (in second) to achieve alveolar concentration of desflurane 1, 2, 3, 4, 5 and 6% | participants will be followed until alveolar concentration of desflurane reaches 6%, as expected of 15 minutes

SECONDARY OUTCOMES:
Heart rate | participants will be followed until alveolar concentration of desflurane reaches 6%, as expected of 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen, Thailand